CLINICAL TRIAL: NCT06288867
Title: Arthroscopic Labral Repair Versus Debridement In Hip Labral Tears: A Prospective Comparative Study
Brief Title: A 12 Months Prospective Study Comparing Functional Outcome Scores in Hip Arthroscopic Labral Repair Versus Debridement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Karim Atef Salem, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD28/2024
Record Dates: First submitted 2024-02-24; First posted 2024-03-01 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Hip Injuries; Acetabular Labral Tear; Femoro Acetabular Impingement
Keywords: Hip Arthroscopy; Labral Repair; Labral Debridement; Acetabular Labral Tear
MeSH Terms: conditions — Hip Injuries; Femoracetabular Impingement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Labral Repair (Active Comparator): Labral tears will be repaired with suture anchors.
  Interventions: Procedure: Arthroscopic Labral Repair
- Labral Debridement (Active Comparator): Labral Debridement will be done by electrocautery
  Interventions: Procedure: Arthroscopic Labral Debridement

INTERVENTIONS:
Procedure: Arthroscopic Labral Repair — Patients with Hip Labral tears will be treated with labral repair
  Arms: Labral Repair
Procedure: Arthroscopic Labral Debridement — Patients with Hip Labral tears will be treated with labral debridement
  Arms: Labral Debridement

SUMMARY:
This study aims to address hip labral tears and compare between arthroscopic labral repair versus debridement.

DETAILED DESCRIPTION:
Hip arthroscopy will be performed with the patient under general anesthesia. The patient will be placed in supine position, and traction and joint access will be controlled by fluoroscopy. An anterolateral portal and an inferior mid-anterior portal will be used. Any labral, chondral, and/or bony pathology (cam or pincer) will be treated. Labral tears may be debrided or repaired. Labral repairs will be secured with suture anchors.

Patient's functions will be evaluated preoperatively and postoperatively at 1, 3 and 6 months and 1 year and at the last follow-up using the Harris Hip Score (HHS), visual analog score (VAS), Hip Outcome Score Activities-Daily Living Subscale (HOS-ADL), and Sport-Specific Subscale (HOS-SSS).

ELIGIBILITY:
Inclusion Criteria:

* Sex: both sexes.
* Age: 18 years - 60 years.
* Femoroacetabular impingement (FAI) including all types (cam, pincer, and combined).
* Traumatic Labral tears

Exclusion Criteria:

* Previous hip surgery.
* Hip joint dysplasia, defined by both center edge (CE) angles <25 degrees and Acetabular Index angle >10 degrees.
* Osteoarthritis grade >2 according to Tönnis classification.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Hip Function, as measured by Hip Outcome Score (HOS) | Baseline, 1 year
  The HOS is a patient-completed measure that consists of an "Activities of Daily Living" subscale (17 scored items) and a "Sports" subscale (9 scored items) in which the response options are presented as 5-point Likert scales (Scores 0-4). Scores for each subscale range from 0% (least function) to 100% (most function).The highest potential score is 68, a higher score represents a higher level of physical function for both the ADL and sports subscales
Change from baseline in Hip Function, as measured by Harris Hip Score (HHS) | Baseline, 1 year
  <70 (poor result), 70-79 (fair result), 80-89 (good result) and >90 (excellent result)
Change from baseline in Pain, as measured by the Visual Analogue Scale (VAS) | Baseline, 1 year
  Scores are measured on a 100 mm VAS. The VAS ranges from 0 to 100 with 0 indicating no pain, and higher scores indicating greater pain

CONTACTS AND LOCATIONS:
Overall Officials: Karim A Salem, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt